CLINICAL TRIAL: NCT01691521
Title: MEA115588 A Randomised, Double-blind, Double-dummy, Placebo-controlled, Parallel-group, Multi-centre Study of the Efficacy and Safety of Mepolizumab Adjunctive Therapy in Subjects With Severe Uncontrolled Refractory Asthma
Brief Title: Efficacy and Safety Study of Mepolizumab Adjunctive Therapy in Subjects With Severe Uncontrolled Refractory Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115588
Record Dates: First submitted 2012-09-20; First posted 2012-09-24 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Asthma
Keywords: safety; SB-240563; efficacy; placebo; eosinophils; mepolizumab; Severe refractory asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mepolizumab IV (Experimental): Mepolizumab 75 mg will be administered intravenously approximately every 4 weeks with the last dose at week 32. Subjects in the Mepolizumab IV arm will receive mepolizumab 75 mg intravenously and placebo SC once every 4 weeks with the last dose at Week 28 (total of 8 doses)
  Interventions: Drug: Mepolizumab IV; Drug: SC Placebo
- Mepolizumab SC (Experimental): Subjects in the Mepolizumab SC arm will receive mepolizumab 100 mg SC and placebo IV once every 4 weeks with the last dose at Week 28 (total of 8 doses)
  Interventions: Drug: Mepolizumab SC; Drug: IV Placebo
- Placebo (Placebo Comparator): Subjects in the Placebo arm will receive matching placebo SC and placebo IV once every 4 weeks with the last dose at Week 28 (total of 8 doses)
  Interventions: Drug: IV Placebo; Drug: SC Placebo

INTERVENTIONS:
Drug: Mepolizumab IV — Mepolizumab 75 mg IV will be administered every 4 weeks with the last dose at Week 28
  Arms: Mepolizumab IV
Drug: Mepolizumab SC — Mepolizumab 100 mg SC will be administered every 4 weeks with the last dose at Week 28
  Arms: Mepolizumab SC
Drug: IV Placebo — Normal saline (placebo) will be administered IV every 4 weeks with the last dose at Week 28
  Arms: Mepolizumab SC; Placebo
Drug: SC Placebo — Normal saline (placebo) will be administered SC every 4 weeks with the last dose at Week 28
  Arms: Mepolizumab IV; Placebo

SUMMARY:
This study will evaluate two dose regimens of mepolizumab [75mg intravenous (i.v.) or 100mg subcutaneous (SC) every 4 weeks] compared with placebo over a 32 week treatment period in subjects with severe refractory asthma with elevated blood eosinophils. Efficacy will be measured by a reduction in the frequency of asthma exacerbations. Additional efficacy assessments will include measurements of lung function, symptom scores, and quality of life. Safety will be assessed by clinical laboratory samples, ECGs, immunogenicity and adverse events.

This study is intended to replicate the Phase IIb/III study MEA112997. Subjects in MEA115588, who meet all eligibility criteria at screening visit, will enter the run-in period. Those subjects that are not able/eligible to be randomised at the end of the 6 week run-in period will be deemed run-in failures. Subjects will remain on their current maintenance therapy throughout the run-in, double-blind treatment administration and follow-up periods. Subjects who meet the randomisation eligibility criteria will be randomised in a 1:1:1 ratio to receive one of the following treatments every 4 weeks for a total of 8 doses: Mepolizumab 75 miligram (mg) i.v. and placebo SC, or Mepolizumab 100 mg SC and placebo i.v. or Placebo i.v. and placebo SC.

Subjects that receive all 8 doses of double-blind treatment, and meet the eligibility criteria for the Open-Label Extension (OLE) Study, will be offered the opportunity to participate in the OLE trial.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent prior to participation in the study
* At least 12 years of age at visit 1 and a minimum weight of 45 kilogram (kg)
* A well-documented requirement for regular treatment with high dose inhaled corticosteroid (ICS) in the 12 months prior to Visit 1 with or without maintenance oral corticosteroids (OCS)
* Current treatment with an additional controller medication, besides ICS, for at least 3 months or a documented failure in the past 12 months of an additional controller medication for at least 3 successive months
* Prior documentation of eosinophilic asthma or high likelihood of eosinophilic asthma
* At Visit 1, a pre-bronchodilator FEV1 <80% (for subjects >= 18 years of age), a pre-bronchodilator FEV1 <90% or FEV1:FVC ratio <0.8 (for subjects 12-17 years of age).
* Previously confirmed history of two or more exacerbations requiring treatment with systemic CS
* Male or Eligible Female (females of childbearing potential must commit to consistent and correct use of an acceptable method of birth control)
* French subjects will be included only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Current smokers or former smokers with a smoking history of >=10 pack years
* Presence of a known pre-existing, clinically important lung condition other than asthma
* A current malignancy or previous history of malignancy in less than 12 months
* Known, pre-existing, unstable liver disease cirrhosis and known biliary abnormalities
* Known, pre-existing severe or clinically significant cardiovascular disease
* known, pre-existing other concurrent clinically significant medical conditions that are uncontrolled with standard treatment
* Subjects with any eosinophilic diseases
* QTc(F) ≥450msec or QTc(F) ≥480 msec
* A history of alcohol/substance abuse
* Subject with known immunodeficiency
* Subjects who have received omalizumab within 130 days of Visit 1 or any monoclonal antibody (other than Xolair) to treat inflammatory disease within 5 half-lives of Visit 1
* Subjects who have received treatment with an investigational drug within the past 30 days or five terminal phase half-lives of the drug whichever is longer
* Subjects with allergy/intolerance to a monoclonal antibody or biologic.
* Subjects who are pregnant or breastfeeding
* Subjects who have known evidence of lack of adherence to controller medications and/or ability to follow physician's recommendations
* Previously participated in any study with mepolizumab and received investigational product (including placebo)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2012-10-08; Primary Completion 2014-01-01 (Actual); Study Completion 2014-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (114):
- United States (20):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Albany, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Salt Lake City, Utah
- Argentina (5):
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
- Australia (5):
  - GSK Investigational Site, New Lambton, New South Wales
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
  - GSK Investigational Site, Parkville
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Canada (11):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Chile (3):
  - GSK Investigational Site, Rancagua, Reg Del Libert Bern Ohiggins
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Talcahuano
- France (7):
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Perpignan
  - GSK Investigational Site, Saint-Pierre
- Germany (10):
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (8):
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Pietra Ligure (SV), Liguria
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Perugia, Umbria
  - GSK Investigational Site, Cittadella PD, Veneto
- Japan (13):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Mexico (3):
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, México DF
- Russia (3):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- South Korea (10):
  - GSK Investigational Site, Anyang-si
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Cheongju, Chungcheongbuk-do
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Donggu Gwangju
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju-si, Jeollabuk-Do
  - GSK Investigational Site, Kangwon-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Kyonggi-do
- Spain (3):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
- Ukraine (4):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Mykolayiv
  - GSK Investigational Site, Vinnytsia
- United Kingdom (5):
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, London
  - GSK Investigational Site, Plymouth
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Chen W, Reddel HK, FitzGerald JM, Beasley R, Janson C, Sadatsafavi M. Can we predict who will benefit most from biologics in severe asthma? A post-hoc analysis of two phase 3 trials. Respir Res. 2023 May 2;24(1):120. doi: 10.1186/s12931-023-02409-2. PMID 37131185
- [Derived] Lemiere C, Taille C, Lee JK, Smith SG, Mallett S, Albers FC, Bradford ES, Yancey SW, Liu MC. Impact of baseline clinical asthma characteristics on the response to mepolizumab: a post hoc meta-analysis of two Phase III trials. Respir Res. 2021 Jun 22;22(1):184. doi: 10.1186/s12931-021-01767-z. PMID 34158028
- [Derived] Gibson PG, Prazma CM, Chupp GL, Bradford ES, Forshag M, Mallett SA, Yancey SW, Smith SG, Bel EH. Mepolizumab improves clinical outcomes in patients with severe asthma and comorbid conditions. Respir Res. 2021 Jun 7;22(1):171. doi: 10.1186/s12931-021-01746-4. PMID 34098955
- [Derived] Best N, Price RG, Pouliquen IJ, Keene ON. Assessing efficacy in important subgroups in confirmatory trials: An example using Bayesian dynamic borrowing. Pharm Stat. 2021 May;20(3):551-562. doi: 10.1002/pst.2093. Epub 2021 Jan 21. PMID 33475231
- [Derived] Wardlaw A, Howarth PH, Israel E, Taille C, Quirce S, Mallett S, Bates S, Albers FC, Kwon N. Fungal sensitization and its relationship to mepolizumab response in patients with severe eosinophilic asthma. Clin Exp Allergy. 2020 Jul;50(7):869-872. doi: 10.1111/cea.13680. Epub 2020 Jun 25. No abstract available. PMID 32515118
- [Derived] Kim MK, Park HS, Park CS, Min SJ, Albers FC, Yancey SW, Mayer B, Kwon N. Efficacy and safety of mepolizumab in Korean patients with severe eosinophilic asthma from the DREAM and MENSA studies. Korean J Intern Med. 2021 Mar;36(2):362-370. doi: 10.3904/kjim.2019.198. Epub 2020 May 26. PMID 32450626
- [Derived] Khurana S, Brusselle GG, Bel EH, FitzGerald JM, Masoli M, Korn S, Kato M, Albers FC, Bradford ES, Gilson MJ, Price RG, Humbert M. Long-term Safety and Clinical Benefit of Mepolizumab in Patients With the Most Severe Eosinophilic Asthma: The COSMEX Study. Clin Ther. 2019 Oct;41(10):2041-2056.e5. doi: 10.1016/j.clinthera.2019.07.007. Epub 2019 Aug 22. PMID 31447130
- [Derived] Khurana S, Lyness JM, Mallett S, Nelsen LM, Prazma CM, Albers FC, Forshag M, Llanos JP, Yancey SW, Ortega HG. Association of depressive symptoms with health status and markers of uncontrolled severe asthma. Allergy Asthma Proc. 2019 Jul 1;40(4):230-239. doi: 10.2500/aap.2019.40.4229. PMID 31262378
- [Derived] Nelsen LM, Cockle SM, Gunsoy NB, Jones P, Albers FC, Bradford ES, Mullerova H. Impact of exacerbations on St George's Respiratory Questionnaire score in patients with severe asthma: post hoc analyses of two clinical trials and an observational study. J Asthma. 2020 Sep;57(9):1006-1016. doi: 10.1080/02770903.2019.1630640. Epub 2019 Jun 28. PMID 31251094
- [Derived] Yancey SW, Bradford ES, Keene ON. Disease burden and efficacy of mepolizumab in patients with severe asthma and blood eosinophil counts of >/=150-300 cells/muL. Respir Med. 2019 May;151:139-141. doi: 10.1016/j.rmed.2019.04.008. Epub 2019 Apr 8. PMID 31047111
- [Derived] Ortega HG, Meyer E, Brusselle G, Asano K, Prazma CM, Albers FC, Mallett SA, Yancey SW, Gleich GJ. Update on immunogenicity in severe asthma: Experience with mepolizumab. J Allergy Clin Immunol Pract. 2019 Sep-Oct;7(7):2469-2475.e1. doi: 10.1016/j.jaip.2019.03.042. Epub 2019 Apr 5. No abstract available. PMID 30954640
- [Derived] Ortega H, Menzies-Gow A, Llanos JP, Forshag M, Albers F, Gunsoy N, Bradford ES, Yancey SW, Kraft M. Rapid and Consistent Improvements in Morning PEF in Patients with Severe Eosinophilic Asthma Treated with Mepolizumab. Adv Ther. 2018 Jul;35(7):1059-1068. doi: 10.1007/s12325-018-0727-8. Epub 2018 Jun 15. PMID 29949045
- [Derived] Ortega H, Yancey SW, Keene ON, Gunsoy NB, Albers FC, Howarth PH. Asthma Exacerbations Associated with Lung Function Decline in Patients with Severe Eosinophilic Asthma. J Allergy Clin Immunol Pract. 2018 May-Jun;6(3):980-986.e1. doi: 10.1016/j.jaip.2017.12.019. Epub 2018 Feb 15. PMID 29398640
- [Derived] Gunsoy NB, Cockle SM, Yancey SW, Keene ON, Bradford ES, Albers FC, Pavord ID. Evaluation of Potential Continuation Rules for Mepolizumab Treatment of Severe Eosinophilic Asthma. J Allergy Clin Immunol Pract. 2018 May-Jun;6(3):874-882.e4. doi: 10.1016/j.jaip.2017.11.026. Epub 2017 Dec 16. PMID 29258789
- [Derived] Albers FC, Price RG, Smith SG, Yancey SW. Mepolizumab efficacy in patients with severe eosinophilic asthma receiving different controller therapies. J Allergy Clin Immunol. 2017 Nov;140(5):1464-1466.e4. doi: 10.1016/j.jaci.2017.06.010. Epub 2017 Jul 4. No abstract available. PMID 28687231
- [Derived] Magnan A, Bourdin A, Prazma CM, Albers FC, Price RG, Yancey SW, Ortega H. Treatment response with mepolizumab in severe eosinophilic asthma patients with previous omalizumab treatment. Allergy. 2016 Sep;71(9):1335-44. doi: 10.1111/all.12914. Epub 2016 May 24. PMID 27087007
- [Derived] Ortega HG, Liu MC, Pavord ID, Brusselle GG, FitzGerald JM, Chetta A, Humbert M, Katz LE, Keene ON, Yancey SW, Chanez P; MENSA Investigators. Mepolizumab treatment in patients with severe eosinophilic asthma. N Engl J Med. 2014 Sep 25;371(13):1198-207. doi: 10.1056/NEJMoa1403290. Epub 2014 Sep 8. PMID 25199059
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 115588 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115588 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115588 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115588 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115588 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115588 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115588 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Par. who met the eligibility criteria at screening, entered the Run-in period for a minimum of 1 week and a maximum of 6 weeks. Par. who received all 8 doses and met the eligibility criteria were offered the opportunity to participate in an open label extension (OLE) study. Par. not entering the OLE study completed the Follow-up Visit.
Pre-assignment Details: A total of 802 participants (par.) were screened; 82 were Screen failures; 140 were Run-in failures; 580 were randomized, of which 576 received at least 1 dose of study drug.
Groups:
- Placebo: Participants received placebo intravenously (IV) plus placebo subcutaneously (SC) every 4 weeks (for a total of 8 doses), with the last dose at Week 28. The SC dose and the IV dose were administered into separate arms. A topical anaesthetic was permitted at the injection site to minimize discomfort, as needed. Rescue personnel and rescue medications (salbutamol/albuterol) /equipment were available throughout the study.
- Mepolizumab 75 mg IV: Participants received mepolizumab 75 milligrams (mg) IV plus placebo SC every 4 weeks (for a total of 8 doses), with the last dose at Week 28. The SC dose and the IV dose were administered into separate arms. A topical anaesthetic was permitted at the injection site to minimize discomfort, as needed. Rescue personnel and rescue medications (salbutamol/albuterol) /equipment were available throughout the study.
- Mepolizumab 100 mg SC: Participants received placebo IV plus mepolizumab 100 mg SC every 4 weeks (for a total of 8 doses), with the last dose at Week 28. The SC dose and the IV dose were administered into separate arms. A topical anaesthetic was permitted at the injection site to minimize discomfort, as needed. Rescue personnel and rescue medications (salbutamol/albuterol) /equipment were available throughout the study.
Period: Overall Study
Arm/Group | Placebo | Mepolizumab 75 mg IV | Mepolizumab 100 mg SC
Started | 191 | 191 | 194
Completed | 179 | 175 | 185
Not Completed | 12 | 16 | 9
Not completed — Adverse Event | 4 | 0 | 1
Not completed — Lack of Efficacy | 1 | 1 | 2
Not completed — Protocol Violation | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo IV plus placebo SC every 4 weeks (for a total of 8 doses), with the last dose at Week 28. The SC dose and the IV dose were administered into separate arms. A topical anaesthetic was permitted at the injection site to minimize discomfort, as needed. Rescue personnel and rescue medications (salbutamol/albuterol) /equipment were available throughout the study.
- Mepolizumab 75 mg IV: Participants received mepolizumab 75 mg IV plus placebo SC every 4 weeks (for a total of 8 doses), with the last dose at Week 28. The SC dose and the IV dose were administered into separate arms. A topical anaesthetic was permitted at the injection site to minimize discomfort, as needed. Rescue personnel and rescue medications (salbutamol/albuterol) /equipment were available throughout the study.
- Total: Total of all reporting groups
Arm/Group | Placebo | Mepolizumab 75 mg IV | Mepolizumab 100 mg SC | Total
Number analyzed (Participants) | 191 | 191 | 194 | 576
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.2 (14.26) | 50.0 (14.03) | 51.2 (14.55) | 50.1 (14.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 106 | 116 | 329
  Male | 84 | 85 | 78 | 247
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 3 | 6 | 7 | 16
  American Indian or Alaskan Native | 0 | 0 | 1 | 1
  Asian - Central/South Asian Heritage | 1 | 1 | 0 | 2
  Asian - East Asian Heritage | 15 | 15 | 15 | 45
  Asian - Japanese Heritage | 18 | 17 | 17 | 52
  Asian - South East Asian Heritage | 4 | 0 | 2 | 6
  White - Arabic/North African Heritage | 4 | 3 | 4 | 11
  White - White/Caucasian/European Heritage | 144 | 148 | 148 | 440
  Mixed Race | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Clinically Significant Exacerbations of Asthma Per Year
Description: Clinically significant exacerbations of asthma are defined as worsening of asthma which required use of systemic corticosteroids (IV or oral steroid like prednisone, for at least 3 days or a single intramuscular (IM) corticosteroid (CS) dose is required. For maintenance of systemic corticosteroids, at least double the existing maintenance dose for at least 3 days was required) and/or hospitalization and/or emergency department (ED) visits. The frequency of clinically significant exacerbations of asthma over the 32-week treatment period is expressed as the number of exacerbations per year. Analysis of the number of exacerbations performed using a negative binomial model with covariates of treatment group, baseline maintenance OCS therapy (OCS vs. no OCS), region, exacerbations in the year prior to the study (as an ordinal variable) and baseline % predicted FEV1, and with logarithm of time on treatment as an offset variable.
Time Frame: From randomization (Week 0) to Week 32 or if Early Withdrawal (EW) 4 weeks post last dose
Population: Modified Intent-to-Treat (ITT) Population: all participants who were randomized and who received at least one dose of trial medication. 'Modified' implies that, in cases where there is is a discrepancy between randomized and actual treatment the analysis used the actual treatment received by the participant rather than the randomized treatment.
Measure: Number; unit: Number of exacerbations per year
Arm/Group | Placebo | Mepolizumab 75 mg IV | Mepolizumab 100 mg SC
Number analyzed (Participants) | 191 | 191 | 194
Number of exacerbations per year | 1.74 | 0.93 | 0.83
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 75 mg IV; Test type: Superiority or Other; p < 0.001, Negative binomial model — Hochberg procedure with a gamma parameter of 1 used for multiplicity adjustment; Rate Ratio = 0.53, 95% CI 2-sided [0.40 to 0.72] — Number of exacerbations per year in the mepolizumab 75mg IV arm divided by the number of exacerbations per year in the placebo arm
Statistical Analysis 2: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Superiority or Other; p < 0.001, Negative binomial model — Hochberg procedure with a gamma parameter of 1 used for multiplicity adjustment; Rate Ratio = 0.47, 95% CI 2-sided [0.35 to 0.64] — Number of exacerbations per year in the mepolizumab 100 mg SC arm divided by the number of exacerbations per year in the placebo arm

2. Secondary Outcome: Number of Clinically Significant Exacerbations Requiring Hospitalization (Including Intubation and Admittance to an Intensive Care Unit [ICU]) or ED Visits Per Year
Description: as for outcome 1
Time Frame: From randomization (Week 0) to Week 32 or if Early Withdrawal (EW) 4 weeks post last dose
Population: ITT Population
Measure: Number; unit: Number of exacerbations per year
Arm/Group | Placebo | Mepolizumab 75 mg IV | Mepolizumab 100 mg SC
Number analyzed (Participants) | 191 | 191 | 194
Number of exacerbations per year | 0.20 | 0.14 | 0.08

3. Secondary Outcome: Number of Clinically Significant Exacerbations Requiring Hospitalization (Including Intubation and Admittance to an ICU) Per Year
Description: Clinically significant exacerbations of asthma is defined as worsening of asthma which required use of systemic corticosteroids (IV or oral steroid like prednisone, for at least 3 days or a single intramuscular (IM) corticosteroid (CS) dose is required. For maintenance of systemic corticosteroids, at least double the existing maintenance dose for at least 3 days was required) and/or hospitalization. The frequency of clinically significant exacerbations of asthma over the 32-week treatment period is expressed as the number of exacerbations per year. Analysis of the number of exacerbations performed using a negative binomial model with covariates of treatment group, baseline maintenance OCS therapy (OCS vs. no OCS), region, exacerbations in the year prior to the study (as an ordinal variable) and baseline % predicted FEV1, and with logarithm of time on treatment as an offset variable.
Time Frame: From randomization (Week 0) to Week 32 or if Early Withdrawal (EW) 4 weeks post last dose
Population: ITT Population
Measure: Number; unit: Number of exacerbations per year
Arm/Group | Placebo | Mepolizumab 75 mg IV | Mepolizumab 100 mg SC
Number analyzed (Participants) | 191 | 191 | 194
Number of exacerbations per year | 0.10 | 0.06 | 0.03

4. Secondary Outcome: Mean Change From Baseline in Clinic Pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) at Week 32
Description: FEV1 is defined as the volume of air expelled from the lungs in 1 second. Pre-bronchodilator FEV1 measurements were taken by spirometry. The change from Baseline is defined as the difference between the value of the endpoint at the time point of interest and the baseline value. Analysis performed using mixed model repeated measures with covariates of baseline, region, baseline maintenance OCS therapy (OCS vs. no OCS), exacerbations in the year prior to the study (as an ordinal variable), treatment and visit, plus interaction terms for visit by baseline and visit by treatment group.
Time Frame: Baseline, Week 32
Population: ITT Population. Only participants with a Baseline FEV1 available and at least one post-Baseline FEV1 measurement were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Milliliters (mL)
Arm/Group | Placebo | Mepolizumab 75 mg IV | Mepolizumab 100 mg SC
Number analyzed (Participants) | 189 | 188 | 192
Milliliters (mL) | 86 (31.4) | 186 (31.5) | 183 (31.1)

5. Secondary Outcome: Mean Change From Baseline in the St. George's Respiratory Questionnaire Total Score at Week 32
Description: The St. George's Respiratory Questionnaire is an established instrument, comprising 50 questions, evaluating symptoms, activity, and impacts; to measure Quality of Life in participants with diseases of airway obstruction and to elicit the participant's opinion of his/her health. The lowest possible value is zero and the highest possible value is 100. The higher values correspond to greater impairment in quality of life. The questionnaire was administered at Baseline (Visit 2) and at the Exit Visit (approximately 4 weeks after the last dose of study treatment). The change from baseline is defined as the difference between the value of the endpoint at the time point of interest and the baseline value. Analysis performed using analysis of covariance with covariates of baseline, region, baseline maintenance OCS therapy (OCS vs. no OCS), exacerbations in the year prior to the study (as an ordinal variable), baseline % predicted FEV1, and treatment.
Time Frame: Baseline, Week 32
Population: ITT Population. Note that only participants with a Baseline and Week 32 assessment were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Mepolizumab 75 mg IV | Mepolizumab 100 mg SC
Number analyzed (Participants) | 177 | 174 | 184
Scores on a scale | -9.0 (1.16) | -15.4 (1.16) | -16.0 (1.13)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs were defined as events occurring from the first dose of investigational product until 28 days after the last dose of investigational product, up to 32 weeks.
Description: Serious adverse events (SAEs) and Non-serious AEs were collected in members of Intent-to-Treat (ITT) Population, comprised of all participants who were randomized and who received at least one dose of study medication.
Arm/Group | Placebo | Mepolizumab 75 mg IV | Mepolizumab 100 mg SC
Serious Adverse Events (participants affected / at risk) | 27/191 | 14/191 | 16/194
Other Adverse Events (participants affected / at risk) | 143/191 | 142/191 | 132/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=191) | Mepolizumab 75 mg IV (N=191) | Mepolizumab 100 mg SC (N=194)
Asthma (Respiratory, thoracic and mediastinal disorders) | 14 | 9 | 5
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 2
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Vulval abscess (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0
Inflammation of wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0
Calculus urethral (Renal and urinary disorders) | 1 | 0 | 0
Nephrogenic diabetes insipidus (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Intracranial lipoma (Congenital, familial and genetic disorders) | 1 | 0 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=191) | Mepolizumab 75 mg IV (N=191) | Mepolizumab 100 mg SC (N=194)
Nasopharyngitis (Infections and infestations) | 46 | 45 | 33
Headache (Nervous system disorders) | 33 | 46 | 39
Upper respiratory tract infection (Infections and infestations) | 27 | 22 | 24
Sinusitis (Infections and infestations) | 18 | 11 | 18
Bronchitis (Infections and infestations) | 16 | 14 | 9
Asthma (Respiratory, thoracic and mediastinal disorders) | 16 | 11 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 12 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 11 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 10 | 11
Injection site reaction (General disorders) | 6 | 5 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 5
Fatigue (General disorders) | 9 | 8 | 5
Gastroenteritis (Infections and infestations) | 6 | 10 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 3 | 8
Diarrhoea (Gastrointestinal disorders) | 11 | 4 | 5
Influenza (Infections and infestations) | 6 | 10 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 7 | 7
Dizziness (Nervous system disorders) | 8 | 4 | 6
Nausea (Gastrointestinal disorders) | 8 | 4 | 5
Urinary tract infection (Infections and infestations) | 2 | 5 | 8
Pharyngitis (Infections and infestations) | 3 | 5 | 6
Eczema (Skin and subcutaneous tissue disorders) | 2 | 2 | 9
Hypertension (Vascular disorders) | 4 | 6 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2 | 7
Migraine (Nervous system disorders) | 6 | 1 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 3
Rhinitis (Infections and infestations) | 4 | 7 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 2
Hypersensitivity (Immune system disorders) | 3 | 6 | 2
Toothache (Gastrointestinal disorders) | 3 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.